CLINICAL TRIAL: NCT04905589
Title: Effect of Combined Intake of Medium Chain Triglycerides (MCT) At Breakfast and Whey Protein Isolate (WPI) Preload At Lunch and Dinner on Diurnal Glucose and Satiety
Brief Title: Medium Chain Triglycerides (MCT) and Whey Protein Isolate (WPI) for Type 2 Diabetes Patients (Combine)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 19.18.CLI
Record Dates: First submitted 2021-05-12; First posted 2021-05-27 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Open-label - randomization-concealed trial randomized in a 1:1:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ARM A (Placebo Comparator): Subsequent order of intake :
  Iso-voluminous water, breakfast, iso-voluminous water, lunch, iso-voluminous water, dinner
  Interventions: Other: Iso-voluminous water
- ARM B (Active Comparator): Subsequent order of intake :
  MCT in liquid form (75 ml of BetaQuik™), breakfast, iso-voluminous water, lunch, iso-voluminous water, dinner
  Interventions: Dietary Supplement: BetaQuik™; Other: Iso-voluminous water
- ARM C (Active Comparator): Subsequent order of intake:
  MCT in liquid form (75 ml of BetaQuik™), breakfast, WPI in liquid from (12.5g of WheyBasics in 200ml water), lunch, WPI in liquid from (12.5g of WheyBasics in 200ml water)), dinner
  Interventions: Dietary Supplement: BetaQuik™; Dietary Supplement: WheyBasics

INTERVENTIONS:
Dietary Supplement: BetaQuik™ — MCT (Medium chain triglycerides)
  Arms: ARM B; ARM C
Dietary Supplement: WheyBasics — Whey Protein Isolate
  Arms: ARM C
Other: Iso-voluminous water — Iso-voluminous Water as comparitor to Betaquik or WheyBasics
  Arms: ARM A; ARM B

SUMMARY:
Evaluation of effect on diurnal glycaemia following consumption of MCT and whey protein in patients with type 2 diabetes

DETAILED DESCRIPTION:
The purpose of this study (Combine) is to evaluate the effects of Combined Intake of Medium chain triglycerides (MCT) at breakfast and whey protein isolate (WPI) preload at lunch and dinner for patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 25 to 65 years of age, inclusive.
2. Subjects with a BMI of ≤ 40kg/m2.
3. Established diagnosis of Type 2 diabetes mellitus (T2DM), documented by either HbA1c 6.5 -10.0% or active therapy with metformin at a daily dose of up to 3000 mg at screening.
4. Willing and able to sign written informed consent prior to study entry.
5. Subjects with laboratory parameters within normal range, or showing no clinically relevant deviations, as judged by the investigator.
6. Willing and able to comply with the requirements of the study protocol.

Exclusion Criteria:

1. Fasting blood glucose >11mmol/L at screening.
2. Elevated liver transaminases > 3 Upper limit of normal at screening.
3. Ongoing or recent (i.e. < 3month) insulin therapy.
4. Ongoing or recent (i.e. < 3month) GLP-1 therapy.
5. Ongoing or recent (i.e. < 3month) treatment with any oral or injectable glucose-lowering drug other than metformin.
6. Ongoing or recent weight loss interventions (e.g. dietary weight loss programmes) or any history of bariatric surgery.
7. Ongoing treatment with anorectic drugs, steroids, medications known to affect gastric motility, or any condition known to affect gastro-intestinal integrity and food absorption.
8. Major medical/surgical event requiring hospitalization in the last 3 months.
9. Known allergy and intolerance to product components.
10. Alcohol intake higher than 4 units per day in line with National Health Service guidelines.
11. History of regular smoking (daily or most days in a week) or use of nicotine products (3 or more nicotine containing products).
12. Have a hierarchical link with the research team members.
13. Subjects who have been dosed in another clinical trial with any investigational drug/new chemical entity within 3 months or 5 half-lives (whichever is longer) prior to screening, or subjects currently participating in any investigational trial.
14. Positive pregnancy test at screening for women of child-bearing potential.
15. Subject who, in the judgment of the investigator, is likely to be noncompliant or uncooperative during the study due to language barrier, poor mental development or any other reason.
16. Subjects with fasting blood glucose that is not within 20% of the value at the previous study visit. Note: In such cases, subjects can come in on another day within the visit window at the discretion of the investigator, however, subjects will be discontinued if the same observation is made at the new visit.
17. Evidence of eating disorders and regularly skipping breakfast and dinner.
18. Current or recent history (in last 3 months) of clinically significant gastrointestinal, liver, cardiovascular, clotting, metabolic or endocrine disorders, apart from T2DM, that in the opinion of the investigator might put the subject at risk by entering the study or interfere with the aims of the study.
19. Total score of ≥ 20 on the Eating Attitude Test (EAT-26) at the screening visit.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Diurnal glucose Incremental area under curve (iAUC) concentrations | 115 days
  Constant glucose monitoring (CGM) comparing treatment regimen A-B-C

SECONDARY OUTCOMES:
Glucose concentrations | 115 days
  Mean, standard deviation and coefficient of variation of 24h glucose concentration as 24h 24h assessed by CGM
Area under curve (AUC) glucose | 115 days
  24h assessed by CGM
Incremental area under curve (iAUC) glucose | 115 days
  24h assessed by CGM
Visual Analogue Scale (VAS) questionnaire | 115 days
  100-point VAS on satiety
Glucose mean | 115 days
  Arterialised blood concentration
Glucose Incremental area under curve (iAUC) | 115 days
  Arterialised blood concentration
Leptin mean | 115 days
  Arterialised blood concentration
Leptin Incremental area under curve (iAUC) | 115 days
  Arterialised blood concentration
Gastric inhibitory polypeptide (GIP) - GLP-1 mean | 115 days
  Arterialised blood concentration
Glucagon-like peptide-1 (GLP-1) mean | 115 days
  Arterialised blood concentration
Gastric inhibitory polypeptide (GIP) - Incremental area under curve (iAUC) | 115 days
  Arterialised blood concentration
Glucagon-like peptide-1 (GLP-1) Incremental area under curve (iAUC) | 115 days
  Arterialised blood concentration
Peptide tyrosine tyrosine (PYY) mean | 115 days
  Arterialised blood concentration
Peptide tyrosine tyrosine (PYY) Incremental area under curve (iAUC) | 115 days
  Arterialised blood concentration

CONTACTS AND LOCATIONS:
Overall Officials: Professor Kostas Tsintzas, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pabla P, Mallinson J, Nixon A, Keeton M, Cooper S, Marshall M, Jacques M, Brown S, Johansen OE, Cuenoud B, Karagounis LG, Tsintzas K. Effect of medium-chain triglycerides and whey protein isolate preloads on glycaemia in type 2 diabetes: a randomized crossover study. Am J Clin Nutr. 2025 Feb;121(2):232-245. doi: 10.1016/j.ajcnut.2024.12.022. Epub 2024 Dec 26. PMID 39732398